CLINICAL TRIAL: NCT01963403
Title: Relief of Bleeding on the Implant: Treatment of Unacceptable Bleeding Patterns in ETG Implant Users With a Combined Oral Contraceptive: A Placebo-Controlled Randomized Trial
Brief Title: Treatment of Unacceptable Bleeding Patterns in ETG Implant Users With an Oral Contraceptive
Acronym: ROBI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Futility of recruitment
Sponsor: University of California, Davis (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Mitchell Creinin, MD, Professor and Director of Family Planning, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 478388; MISP 50618 (Other Grant/Funding Number: Merck Sharp & Dohme Corp.)
Record Dates: First submitted 2013-10-10; First posted 2013-10-16 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Abnormal Uterine Bleeding, Unspecified; Uterine Bleeding Heavy
Keywords: etonogestrel implant; birth control; irregular bleeding; heavy bleeding
MeSH Terms: conditions — Metrorrhagia | interventions — Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EE 30mcg/LNG 150mcg (Active Comparator): combined oral contraceptive pill: ethinyl estradiol (EE) 30mcg/levonorgestrel 150mcg); 1 pill per day; daily during study participation (up to 84 days)
  Interventions: Drug: EE 30mcg/LNG 150mcg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EE 30mcg/LNG 150mcg — 1 pill per day; daily during study participation (up to 84 days)
  Other Names: Levlen28; Levora; Portia 28; Altavera
  Arms: EE 30mcg/LNG 150mcg
Drug: Placebo — 1 pill per day; daily during study participation (up to 84 days)
  Arms: Placebo

SUMMARY:
This double-blinded, placebo-controlled, randomized trial will compare the effects of the use of a combined oral contraceptive pill to a placebo pill for women who are experiencing irregular and/or heavy bleeding associated with the use of an etonogestrel (ETG) implant.

The hypothesis of the study is:

* Use of combined oral contraceptive will significantly improve bleeding patterns for users of ETG implant
* Continuation rate of ETG implant users will be increased by use of combined oral contraceptive in women desiring ETG implant removal because of the undesirable bleeding
* Adverse events will be uncommon and acceptable to women who use a combined oral contraceptive with the ETG implant

DETAILED DESCRIPTION:
Women who are experiencing irregular and/or heavy bleeding associated with the use of an etonogestrel (ETG) implant will be recruited for this study. Women who have bothersome bleeding will be randomized to use either a combined oral contraceptive pill or a placebo pill.

Participants will take one pill every day and record their bleeding patterns on a daily diary.

Participants will have one screening/enrollment visit, two in-person follow up visits, and one telephone follow up contact. Subjects will be enrolled for a total of 84 days (three months).

Participants will be assigned to a treatment group at her screening/enrollment visit. Her first follow up visit will occur 22-28 days after her enrollment. Participants can choose to:

* Continue use of assigned treatment medication
* Discontinue use of assigned treatment medication, but use an open-label combined oral contraceptive pill
* Discontinue the use of assigned treatment medication, decline use of an open-label combined oral contraceptive pill
* Discontinue use of ETG implant.

Participants who choose to continue use of ETG implant will have a follow up telephone contact 50-56 days after her enrollment visit. A final in-person visit will occur 78-84 days after enrollment. Bleeding patterns will be assessed by daily bleeding diaries completed by the participant.

ELIGIBILITY:
Inclusion Criteria:

* Women who have an ETG implant in place
* Women who subjectively experience the side effect of an undesirable bleeding profile such as bleeding irregularity or heavy flow after ETG implant was placed and who desire intervention for this side effect by either treatment of bleeding or removal of the implant
* Age 14 years an older, inclusive

Exclusion Criteria:

* Irregular or heavy bleeding from an etiology other than ETG use (e.g. fibroids, cervical polyp, or other organic cause of bleeding)
* Has attempted prescription treatment for menstrual side effects while using ETG implant
* Has one or more of the conditions considered Category 3 (risks outweigh benefits) or Category 4 (unacceptable health risk) for estrogen-containing oral contraceptives by the Center for Disease Control Medical Eligibility Criteria for Contraceptive Use:

  * Current or history of heart or vascular diseases, including deep venous thrombosis, pulmonary embolism, known thrombogenic mutations, peripartum cardiomyopathy, and complicated valvular heart disease
  * Hypertension, even if adequately controlled
  * Diabetes with vascular involvement
  * Headaches with focal aura, or migraines in women age 35 and older even without focal aura
  * Major surgery with prolonged immobilization
  * Breast cancer (current or past)
  * Severe (decompensated) cirrhosis
  * Acute or flare viral hepatitis
  * Breastfeeding less than 1 month postpartum
  * Post-partum less than 3 weeks
  * 35 years of age and older and smoking
  * Multiple risk factors for arterial cardiovascular disease
  * Systemic Lupus Erythematosus with positive or unknown antiphospholipid antibodies
  * Current symptomatic gallbladder disease or history of cholestasis related to past combined oral contraceptive use
  * On certain anticonvulsants (phenytoin, carbamazepine, barbiturates, primidone, topiramate, oxcarbazepine, lamotrigine)
  * On Ritonavir-boosted protease inhibitors for antiretroviral therapy
* Issues or concerns, in the judgment of the investigator, that may compromise the safety of the subject, impact the subject's adherence to the protocol requirements, or confound the reliability of the data acquired in this study

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Creinin, MD, Principal Investigator — University of California, Davis; Melody Hou, MD, Study Director — University of California, Davis
Locations (2):
- United States (2):
  - University of California, Davis Department of Obstetrics and Gynecology, Sacramento, California
  - Washington University School of Medicine, Department of Obstetrics and Gynecology, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hou MY, McNicholas C, Creinin MD. Combined oral contraceptive treatment for bleeding complaints with the etonogestrel contraceptive implant: a randomised controlled trial. Eur J Contracept Reprod Health Care. 2016 Oct;21(5):361-6. doi: 10.1080/13625187.2016.1210122. Epub 2016 Jul 15. PMID 27419258

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EE 30mcg/LNG 150mcg | Placebo
Started | 13 | 13
Completed | 11 (Follow-up over three months) | 9 (Follow-up over three months)
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 2 | 3
Not completed — Implant removal | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EE 30mcg/LNG 150mcg | Placebo | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.4 (3.8) | 25.8 (5.0) | 25.6 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 13 | 25
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 4 | 3 | 7
  White | 5 | 5 | 10
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26
Primary reason for implant [Count of Participants; unit: Participants]
  Contraception | 11 | 12 | 23
  Bleeding Problem | 1 | 1 | 2
  Dysmenorrhea | 1 | 0 | 1
Duration of implant use [Median (Full Range); unit: days] | 343 [25 to 764] | 109 [41 to 518] | 144.5 [25 to 764]
intervention requested before enrollment [Count of Participants; unit: Participants]
  implant removal | 2 | 3 | 5
  Hormonal treatment | 6 | 4 | 10
  'Some treatment' | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Bleeding Improvement
Description: Bleeding improvement will be measured by participant response to the question of whether she feels her bleeding is improved and she is satisfied with the treatment.
Time Frame: Bleeding improvement will be evaluated during first cycle of study treatment (28 days)
Population: 1 person in each group LTFU at one month, which was the primary outcome
Measure: Count of Participants; unit: Participants
Arm/Group | EE 30mcg/LNG 150mcg | Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Significant improvement | 11 | 5
  Slight improvement | 1 | 3
  No change | 0 | 2
  Slightly worse | 0 | 2
  Significantly worse | 0 | 0

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Participants will be evaluated for adverse events while using a combined oral contraceptive with ETG implant.
Time Frame: Adverse events will be evaluated at each contact (visits at 1 and 3 months, phone contact at 2 months) with the participant
Population: Outcomes at one month; 1 person LTFU at one month in each group
Measure: Count of Participants; unit: Participants
Arm/Group | EE 30mcg/LNG 150mcg | Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Headache | 5 | 4
  Nausea/vomiting | 1 | 1
  Cramping | 0 | 2
  Mood change | 0 | 1
  None of above | 6 | 4

3. Other Pre Specified Outcome: Number of Participants withTreatment Success or Failure
Description: Treatment success will be measured by desire to continue treatment because the initial treatment made the bleeding better.
  Partial failure of the study treatment will be measured by the desire to continue treatment because the initial treatment did not work
  Complete failure of treatment will be measured by the desire to:
  * discontinue treatment because it did not work; no further treatment requested
  * ETG implant removal
  * Desire to use non-study treatment
Time Frame: Evaluated at follow up visits at 1 month and, if subject continues after 1st month, again at 3 months
Population: one month evaluation; 1 subject LTFU at one month in each group
Measure: Count of Participants; unit: Participants
Arm/Group | EE 30mcg/LNG 150mcg | Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Continued assigned treatment | 8 | 5
  Desired COC prescription | 4 | 4
  Desired no treatment | 0 | 2
  Implant removal | 0 | 1

4. Other Pre Specified Outcome: Bleeding Patterns and Number of Participants With Bleeding Improvement
Description: * Bleeding improvement in women who received placebo but opted for open-label treatment after first cycle
  * Bleeding improvement over the 84 days of study participation
  * Bleeding patterns in placebo vs. combined oral contraceptive users
Time Frame: Evaluated at follow up visits at 1 month and, if subject continues after 1st month, again at 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Used COC at Any Time During 3 Months | No Use of COC at Any Time During 3 Months
Number analyzed (Participants) | 16 | 5
Participants
  Bleeding improvement | 12 | 5
  No bleeding improvement | 4 | 0

ADVERSE EVENTS:
Time Frame: Up to 84 days on either medication or placebo.
Description: Adverse events for the drug arms reported combined arms. Placebo adverse events are reported for the single arm.
Arm/Group | EE 30mcg/LNG 150mcg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 6/12 | 8/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EE 30mcg/LNG 150mcg (N=12) | Placebo (N=12)
Headache (General disorders) | 5 (5) | 4 (4)
Nausea/vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cramping (General disorders) | 0 (0) | 2 (2)
Mood change (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No